CLINICAL TRIAL: NCT00591318
Title: IV Ceftriaxone for Refractory Psychosis: a Controlled Trial
Brief Title: A Placebo-controlled Efficacy Study of IV Ceftriaxone for Refractory Psychosis
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study was terminated after enrolling 12 patients due to poor enrollment rates
Sponsor: Research Foundation for Mental Hygiene, Inc. (Other)
Collaborators: National Alliance for Research on Schizophrenia and Depression (Other); New York State Psychiatric Institute (Other)
Responsible Party: Principal Investigator, Brian A Fallon, Professor of Clinical Psychiatry, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 5418
Record Dates: First submitted 2007-12-26; First posted 2008-01-11 (Estimated); Results first posted 2022-01-12 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-11

CONDITIONS: Psychosis; Schizophrenia; Schizoaffective Disorder
Keywords: Ceftriaxone; Psychosis; Schizophrenia; Schizoaffective Disorder
MeSH Terms: conditions — Psychotic Disorders; Schizophrenia | interventions — Ceftriaxone; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- IV Ceftriaxone (Experimental): IV Ceftriaxone 2 grams/day
  Interventions: Drug: ceftriaxone
- IV Placebo (Placebo Comparator): IV Placebo (Normal Saline)
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: ceftriaxone — 2 grams of ceftriaxone given daily, Monday to Friday, excluding major holidays, for a total of 40 doses
  Other Names: "Rocephin"
  Arms: IV Ceftriaxone
Drug: Normal Saline — 50 cc of normal saline, daily, Monday through Friday, except for major holidays, for a total of 40 normal saline infusions.
  Other Names: placebo
  Arms: IV Placebo

SUMMARY:
Many patients with schizophrenia and schizoaffective disorder have symptoms that persist, including hallucinations or delusions, despite adequate pharmacotherapy with antipsychotic drug. Glutamate is a major excitatory neurotransmitter in the brain that has been implicated in several brain diseases. NMDA antagonist drugs cause symptoms of psychosis in otherwise normal persons. It is postulated that reduced NMDA receptor mediated neurotransmission leads to an increase in synaptic glutamate. Excessive synaptic concentrations of glutamate can produce excitatory neurotoxicity. Agents which reduce excess glutamate activity are neuroprotective. This therapeutic strategy has been applied to schizophrenia through the use of compounds that reduce presynaptic release of glutamate or otherwise decrease excessive postsynaptic stimulation, including lamotrigine, memantine and a m-GLU-R2 agonist (LY354740) with the hypothesized result of a reduction in psychotic symptoms.

Recently it was shown that a commonly available antibiotic (ceftriaxone) has the unique neuroprotective function of decreasing the amount of extracellular glutamate in nervous system tissue by increasing the number of glutamate transporter proteins. Our clinical experience with patients who have refractory psychosis and past Lyme disease indicates that in some patients psychosis may improve with IV ceftriaxone therapy. Whether this improvement was due to its antimicrobial or glutamate effect or a placebo effect is uncertain. In a placebo-controlled design, this study investigates the ability of ceftriaxone to decrease psychotic symptoms in patients with refractory psychotic disorders. In addition, the study will examine glutamatergic functional activity before and after treatment using brain imaging with magnetic resonance spectroscopy.

DETAILED DESCRIPTION:
Patients will be screened over the telephone. Information will be gathered from the mental health treatment team and the patient. Most patients who come to this study have had an inadequate or insufficient improvement with clozapine. Upon arrival at the NYS Psychiatric Institute, they review and sign consent to make sure the details of the research study are understood. Comprehensive assessments are conducted, including neurocognitive testing, prior to treatment onset. The treatment is randomized so patients will either receive IV ceftriaxone or IV placebo. Treatment is given Monday through Friday to enable the patient to have weekends off without a plastic tube (angiocath) in the vein of the arm. If after 6 weeks the patient's symptoms are not at least mildly improved, then the treatment will be stopped. If however there are signs of improvement, the treatment will be continued another 2 weeks. If at the end of the "double-blind" part of the study a patient learns he/she received placebo and wishes to be given ceftriaxone, we will provide 4 weeks of ceftriaxone for those patients. The inpatient unit is located in the NYS Psychiatric Institute which is adjacent to the Columbia Medical Center in northern Manhattan. Our new building for the NYS Psychiatric Institute is about 10 years old so the inpatient unit is quite attractive with beautiful views of the Hudson River and the Palisades. There is no financial cost for the inpatient stay nor is there a financial cost for participating in this study.

Patients or family members wishing to learn more about this research study should call 212-543-6510 for more information or call Dr. Fallon directly at 212-543-5487.

ELIGIBILITY:
Inclusion Criteria:

1. Adult age 18-55 (Self Report)
2. Persistent positive symptoms of psychosis despite at least three adequate trials of anti-psychotics as defined by the Texas medical Algorithm Project - one of which is clozapine unless there is a contra-indication. (Review of medical records and conversation with prior treating psychiatrist).
3. Significant positive symptoms, including delusions and/or hallucinations. (Clinical evaluation/interview)
4. Diagnosis of schizophrenia or schizoaffective disorder (DSM-IV Diagnostic Checklist)
5. Patients will be on a stable dose of antipsychotic medication for at least 8 weeks prior to randomization or 4 months if Clozaril (Clinical evaluation)
6. Negative Urine Toxicology (Urine collection at the time of initial evaluation)
7. Patients on other antidepressants/mood stabilizers (except PRN benzodiazepines) will be at the same dose for at least 2 months prior to starting this trial. (Clinical evaluation & record review.)
8. Patient's current treatment has been optimized (Review of medical records and conversation with treating psychiatrist)
9. Patient is likely to tolerate the departure from clinical management required of study participants (Review of medical records and conversation with treating psychiatrist)
10. There is no significant risk of self-injury or violence based on recent history and current mental state (Review of medical records and conversation with treating psychiatrist) -

Exclusion Criteria:

1. Penicillin or cephalosporin allergy (Self-report)
2. Agitation such that patient is likely to be unable to tolerate having an IV line in place.(Behavioral Observation)
3. Current Lyme disease that has not been treated previously. Current or history of liver, kidney, or gall bladder disease or elevated liver function test, elevated BUN over/Cr at screening. Unstable medical illness. History of gall stones (without subsequent cholecystectomy), hypereosinophilic syndrome, sickle cell disease, immunodeficiency or blood clotting disorder. History of inflammatory bowel disease, colon cancer, or C.difficile colitis. (Review of medical history, screening blood test).
4. Inability to be an inpatient for at least 8 weeks. (Discussion with patient (& family if indicated))
5. A history of IV drug abuse. (Review of medical history)
6. Inability to provide informed consent. (Capacity will be assessed by a clinical MD.)
7. Patients who had received IV antibiotic therapy within the last year (Review of medical history)
8. Pregnancy or lactation. For females of child bearing age, the pregnancy test is performed pre-randomization. Since this test cannot detect the very early stage of pregnancy (10 day period between fertilization and implantation), an effective birth control method or sexual abstinence is required during the 15 days before the MR scan and randomization. (Interview & urine pregnancy test pre-randomization)
9. For subjects participating in the MRSpectroscopy component: Current or past history of claustrophobia (Interview and history)
10. For subjects participating in the MRSpectroscopy component Metal implants or paramagnetic objects contained within the body which may pose a risk to the subject or interfere with the MR scan, as determined in consultation with a neuroradiologist and according to the guidelines set forth in the following reference book commonly used by neuroradiologists: "Guide to MR procedures and metallic objects", F.G. Shellock, Lippincott Williams and Wilkins, NY 2001. (Interview and history)
11. History of self-injurious behaviour or other behaviour that might complicate the insertion and maintenance of an angiocath, in the past 2 years (Interview and History)
12. Patient is currently taking Cyclosporine (Interview and Medical records review)

    -

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2007-10-10 (Actual); Primary Completion 2011-03-02 (Actual); Study Completion 2011-03-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian A Fallon, MD, Principal Investigator — New York State Psychiatric Institute
Locations (1):
- NYS Psychiatric Institute, New York, New York, United States

REFERENCES:
- [Background] Rothstein JD, Patel S, Regan MR, Haenggeli C, Huang YH, Bergles DE, Jin L, Dykes Hoberg M, Vidensky S, Chung DS, Toan SV, Bruijn LI, Su ZZ, Gupta P, Fisher PB. Beta-lactam antibiotics offer neuroprotection by increasing glutamate transporter expression. Nature. 2005 Jan 6;433(7021):73-7. doi: 10.1038/nature03180. PMID 15635412

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There were 12 people who signed consent but 2 opted not to start treatment and therefore are not included in the demographics or the treatment results report
Period: Overall Study
Arm/Group | IV Ceftriaxone | IV Placebo
Started | 5 | 5
Completed | 1 (For our protocol, participants in both treatment arms were considered completers if they completed at least 6 weeks. At the 6 week point, if response on PANS was not sufficient (15% or greater), they were considered unlikely to respond and therefore were not given the option of the 2 additional weeks of ceftriaxone or placebo. For the analysis, we used the last observed rating between baseline to week 8 for each participant, regardless of whether the participant completed the study treatments.) | 5 (For our protocol, participants in both treatment arms were considered completers if they completed at least 6 weeks. At the 6 week point, if response on PANS was not sufficient (15% or greater), they were considered unlikely to respond and therefore were not given the option of the 2 additional weeks of ceftriaxone or placebo. For the analysis, we used the last observed rating between baseline to week 8 for each participant regardless of whether the participant completed the study treatments..)
Not Completed | 4 | 0
Not completed — Lack of Efficacy | 2 | 0
Not completed — Adverse Event | 2 | 0

BASELINE CHARACTERISTICS:
Population: We had 12 who signed consent but 2 chose not to enter the treatment component of the study and so our sample size total is 10 for the treatment study
Groups:
- Ceftriaxone: Ceftriaxone Group (n=5)
- Placebo: Placebo Group (n=5)
- Total: Total of all reporting groups
Arm/Group | Ceftriaxone | Placebo | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 41 (12.5) | 38.6 (11.7) | 40.5 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 3 | 4 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 5 | 10
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 3 | 4 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
PANSS Positive [Mean (Standard Deviation); unit: score on a scale] | 16.7 (4.9) | 18.2 (4.9) | 17.3 (4.8)

OUTCOME MEASURES:

1. Primary Outcome: Positive and Negative Syndrome Scale - Positive Subscale
Description: Positive and Negative Syndrome Scale (PANSS) - 7 point scale where 1 is absent and 7 is extreme The positive scale has 7 items. Altogether there are 7 items for the total score (range is a minimum of 7 to a maximum of 49). Lower scores indicate better health.
  We report the Positive scale
Time Frame: Last observation assessed occurring from baseline through to the end of week 8
Population: We included all 10 people who started treatment. We used the last observation carried forward in the final analysis which included all time points from baseline through to the end of week 8.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Ceftriaxone Arm Results: This group was randomized to 2 gms of ceftriaxone given 5 days/week for 8 weeks. If participants were not at least 15% improved at 6 weeks, they were considered unlikely to respond and rated as having completed the randomized phase of treatment.
- Placebo Arm Results: This group was randomized to receive saline given 5 days/week for 8 weeks
Arm/Group | Ceftriaxone Arm Results | Placebo Arm Results
Number analyzed (Participants) | 5 | 5
score on a scale | 17.6 (4.9) | 18.6 (4.3)

2. Secondary Outcome: Scale for the Assessment of Positive Symptoms
Description: Scale evaluates positive symptoms of psychosis rated on a scale of 0-5 for each of the 34 items (0 for absent and 5 for severe).
  Minimum score is 0 and the maximum score is 170; higher scores are worse.
Time Frame: Last observation assessed occurring from baseline through to the end of week 8
Population: All 9 participants had ratings on this scale which were used for the results below. One placebo participant (the missing one of the 10) only had a rating at baseline and so was not included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Ceftriaxone: Group randomized to Ceftriaxone
- Placebo: This group received IV saline
Arm/Group | Ceftriaxone | Placebo
Number analyzed (Participants) | 5 | 4
score on a scale | 27.8 (15.1) | 22.7 (7.9)

3. Secondary Outcome: Hamilton Depression Scale
Description: This is a clinician-administered scale of depression severity with 17 items with scores ranging from 0-7 with higher scores indicating greater severity of depression.
  The range is 0-119, where higher scores indicate greater depression
Time Frame: Last observation assessed occurring from baseline through to the end of week 8
Population: 5 in the ceftriaxone group and 4 in the placebo group had ratings on this scale
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Ceftriaxone: Sample randomized to IV Ceftriaxone
- Placebo: Participants received IV saline
Arm/Group | Ceftriaxone | Placebo
Number analyzed (Participants) | 5 | 4
score on a scale | 15.4 (12.7) | 7.7 (5.5)

4. Secondary Outcome: Hamilton Anxiety Rating Scale
Description: The Hamilton Anxiety Rating Scale is a clinician-administered scale of 14 items, with each item rated 0-4 where 4 is the most severe.
  The range is 0-56 where the higher values indicate greater anxiety.
Time Frame: Last observation assessed occurring from baseline through to the end of week 8
Population: Results from the analysis of data on all 10 participants are presented below
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ceftriaxone | Placebo
Number analyzed (Participants) | 5 | 5
score on a scale | 6.2 (5.4) | 5.8 (2.2)

ADVERSE EVENTS:
Time Frame: Adverse events are reported that occurred during the time period of each participants receipt of randomized treatment (ranging to a maximum of 8 weeks)
Groups:
- Ceftriaxone: Participants randomized to Ceftriaxone
- Saline: Participants randomized to saline
Arm/Group | Ceftriaxone | Saline
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 1/5 | 0/5
Other Adverse Events (participants affected / at risk) | 4/5 | 1/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ceftriaxone (N=5) | Saline (N=5)
Prolongation of hospitalization (Psychiatric disorders) | 1 (1) | 0 (0) — Individual's psychosis symptoms worsened
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ceftriaxone (N=5) | Saline (N=5)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) — Rash on skin that resolved
Diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0) — Diarrhea not due to C.Difficile
Pain (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Pain at site of IV catheter

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No